CLINICAL TRIAL: NCT00344994
Title: An Open-Label Prospective Study of Restless Legs Patients Switched to Ropinirole From Pramipexole to Help Determine the Equipotent Dose
Brief Title: SWITCH:Restless Legs Patients Switched to Ropinirole From Pramipexole
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Dr. Kapil Sethi/ / PI, Georgia Health Sciences University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: gskswitch
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Restless Legs Syndrome
Keywords: Restless Legs Syndrome; Mirapex (pramipexole); Requip(Ropinirole); Dopamine Agonist
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Pramipexole

INTERVENTIONS:
Drug: pramipexole — PO, 0.25mg, 0.50mg, or 0.75mg QHS

SUMMARY:
The purpose of this study is to determine the equipotent dose of ropinirole and pramipexole for patients switched from pramipexole to ropinirole in patients with moderate to severe primary Restless Legs Syndrome (RLS). The rationale behind Switch is that patients with Restless Legs Syndrome can maintain stable efficacy and tolerability if correctly switched from one dopamine agonist to an equipotent dose of another.

DETAILED DESCRIPTION:
BACKGROUND Dopamine agonists such as ropinirole (Requip) and pramipexole (Mirapex) are effective treatments for Restless Legs Syndrome and Parkinson Disease. However, although the safety and efficacy may be established, it is common for clinicians to switch between therapies in order to seek optimal symptomatic relief for their patients. The best strategy for switching from other dopamine agonists to Requip is currently undetermined. Currently, ropinirole is the only medication indicated for the treatment of moderate to severe RLS.

Every patient will have an individual response to each dopamine agonist. Usually patients are switched from one dopamine agonist to another due to the following factors:

* Lack of response or loss of efficacy
* Predictable and dose-related side effects
* Ergot-associated adverse events (pulmonary fibrosis, cardiac valvulopathy, etc.)
* Sleep events (sudden onset of sleep)
* Peripheral edema
* Patient co-morbidities

The lack of clinical data makes it difficult to recommend switching guidelines that are suitable for all patients. It is therefore recommended that the switching regimen be based on clinical judgment with individualization for each patient. Switching from one dopamine agonist to another is dependent upon a number of factors including:

1. The currently prescribed dopamine agonist
2. The dose of the current dopamine agonist
3. Whether dopamine agonist is being administered as monotherapy or as adjunct therapy to L-dopa
4. Individual patient response to both the current agonist and to the other dopamine agonist (efficacy and tolerability)
5. Stage of the disease

In placebo-controlled, clinical trials for Requip, a protocol for switching patients to Requip was not utilized. Patients were generally required to discontinue previous dopamine agonist medications at least two weeks prior to baseline evaluation. Patients already on dopamine agonists were discontinued according to the practices of the investigators.

Methods of switching that have been studied previously include:

1. Withdrawal of the current dopamine agonist according to the manufacturer's recommendations followed by initiation of the other dopamine agonist based upon the manufacturer's recommendations
2. An overnight switch with abrupt cessation of the current dopamine agonist followed by initiation of an estimated equivalent dose of the other dopamine agonist
3. Gradual withdrawal of the current dopamine agonist with simultaneous upward titration of the other dopamine agonist

   STUDY DESIGN

   SWITCH is a principal investigator-initiated, open-label study that is being conducted at two sites, to include the Medical College of Georgia and the VA Medical Center (VAMC). A total of 20 subjects will be enrolled at MCG/VAMC. Individuals who choose to participate will have approximately three to four study visits over a four week time period. Patients with moderate to severe primary Restless Legs Syndrome will be included in the study. All RLS medications will be at a stable dose for at least 4 weeks prior to enrollment. Patients will be switched overnight at the Baseline Visit at a ratio of either 1:4 or 1:6 Mirapex (pramipexole) to Requip (ropinirole) per Conversion Table 1 below:

   Table 1: Conversion Table

   Pramipexole Dose Requip Dose (tablets)

   1:4 conversion

   0.25mg------------------ 1mg (1X1mg)

   0.5mg ------------------ 2mg(1X2mg)

   0.75mg-------------------3mg (1X 3mg)

   1:6 Conversion

   0.25mg------------------1.5mg (3X0.5mg)

   0.5mg ------------------3mg (1X 3mg)

   0.75mg------------------4mg (1X4mg)

   At the baseline study visit, a signed and dated consent will first be obtained from the subject. In addition, inclusion/exclusion criteria will be reviewed before the start of any study procedures.

   During the course of the study, some or all of the following procedures will be performed, when patients come to the clinic for their study visit (Table 2):
   * Health and Medication Review: Ask patients to answer questions about their health, medical history, and their medications. (All visits)
   * Mini-Mental State Examination: Patients will be asked a series of questions to determine their mental status. (Visit 1)
   * CGI-S/CGI-I: (Visits 1, 2, and 4)
   * IRLS: (Visits 1, 2, and 4)
   * Epworth Sleepiness Scale: (Visits 1, 2, and 4)
   * ECG: An "ECG" or "electrocardiogram" is a test that measures the electrical activity of the heart. (Visits 1, 2, and 4)
   * Blood Tests: The study staff will draw about 3 tablespoons. The study doctor will use this blood for Hematology and Chemistry panel laboratory tests. (Visit 1)
   * Pregnancy Tests: If the patient is female and can have children, their blood (about one extra tablespoon will be needed to perform this test) will be tested to see if they are pregnant. Patients will be told if the test results are positive. The results of the test must be negative in order for the patient to be in the study. (Visit 1)
   * Neurological and Physical Exam: The study doctor will perform both a neurological and a physical exam. (Visit 1)
   * Brief Physical Exam (Visits 2 and 4)
   * Concomitant Medication Review (All visits)
   * Blood Pressure, Pulse (Visits 1, 2, and 4)
   * Height (Visit 1)
   * Weight (Visit 1)
   * Study Drug: Give patients a supply of study drug and tell them how to take it. Patients will be asked to bring back all unused study drug to each visit. (Visits 1, 2, and 4)
   * Drug Compliance (Visits 2, 3, and 4)
   * Adverse Event Review (Visits 2, 3, and 4)
   * Telephone Contact: The study doctor or study staff will call the patient to check on his/her health and see how he/she is handling the study drug. If the study doctor decides that the patient is doing well on the medication, Visit 3 could only consist of a telephone contact to include a review of concomitant medications, adverse events, and drug compliance. If the patient is experiencing breakthrough symptoms, a clinic visit will be required for Visit 3.

   All study visits will take approximately two (2) hours and the telephone contact should take no longer than thirty (30) minutes.

   Study Patients will see both the study coordinator and an investigator at every visit.

   At the end of study treatment, subjects will be given treatment options; subjects will have the option of continuing on ropinirole or returning to the use of pramipexole. Subjects will then return to the care of their primary care physician/neurologist.

   USE OF HUMAN SUBJECTS and/or HUMAN DERIVED MATERIALS

   SUBJECT CHARACTERISTICS Patients with moderate to severe Restless Legs Syndrome that are currently taking a stable dose of Pramipexole will be approached during their visit to the MCG Movement Disorders Clinic and the VA Neurology Clinic and asked to participate in SWITCH. If it becomes necessary to recruit from outside of MCG/VAMC, all advertisement materials will be submitted to the HAC for approval prior to use. SWITCH is a double site study. We plan to enroll a total of 25-30 individuals between the two sites. Approximately 20 patients will be enrolled at MCG/VAMC.

   MANAGING SIDE EFFECTS As with all drugs, the possibility of unforeseeable risks and side effects exist. The patients will be told of any important new information that might affect their decision to continue in the study in a timely manner. Their Restless Legs Syndrome may not improve or may worsen, despite participation. In previous studies, patients taking ropinirole reported the following side effects to include: nausea, headache, dizziness, drowsiness, or sleepiness. Individuals taking ropinirole may experience dizziness, nausea, sweaty or faintness when first standing up from lying down. Hallucinations (unreal visions, sounds, or sensations) have also been reported in patients taking ropinirole, especially in elderly patients, patients taking ropinirole with L-dopa, or patients taking higher amounts of ropinirole. If a patient is taking L-dopa for Parkinson's disease, ropinirole may worsen some of the side effects of L-dopa.

   Additionally, ropinirole has been associated with sedating effects, including somnolence and the possibility of falling asleep while engaged in activities of daily living, including operation of a motor vehicle.

   Syncope or symptomatic hypertension may also occur, particularly during initial treatment or dose titration. Patients should be cautioned against rising rapidly after sitting or lying down. Because of possible additive effects, it is recommended that caution be exercised with patients who have sleep disorders or are taking sedating medications, alcohol, CNS depressants, or medications that increase ropinirole plasma levels.

   Patients should get medical help and contact the study doctor or study staff, if they have any of these or any other side effects during the study.

   If the study doctor considers that it is in the patient's best interest to discontinue a current medication so that they can enter the study, the patient may experience some withdrawal symptoms.

   The risks and discomforts of blood drawing from a vein include the possibility of pain or bruising at the site of the blood draw; occasional feelings of lightheadedness; and, rarely, infection at the site of the blood draw.

   Currently, Ropinirole is an FDA approved drug for the treatment of RLS. There are currently other medications used for the treatment of Restless Legs Syndrome such as Pramipexole, gabapentin, Sinemet, clonazepam, opiods (pain medications), benzodiazepines (sleep medications), anticonvulsants (medications to prevent seizures), and iron therapy. The study doctor will discuss the benefits and risks associated with these alternatives with each patient.

   If a research related event arises, the study team will manage the patient's care. In the event of an emergency, the research team is available any time, day or night, via the MCG paging operator.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained
* Males and/or females; females of childbearing potential, who are not currently pregnant, must agree to use a medically accepted method of contraception throughout the study (i.e., oral contraception, intra- uterine device, or a long-acting injectable form of contraception). Barrier methods alone (i.e., condom) are not adequate.
* Age > 18 years to ≤ 80 years
* Patients with moderate to severe primary RLS
* Stable dose of Pramipexole, between 0.25 mg and 0.75mg, for Restless Legs Syndrome for 4 weeks prior to enrollment
* IRLS >15 (before pramipexole was initiated)

Exclusion Criteria:

Anyone who does not fit the criteria stated under "Inclusion Criteria" and anyone who is included in the following criteria:

* Currently taking neuroleptic medications
* Currently taking dopamine blocking anti-emetic medications.
* Currently taking any drug known to substantially inhibit CYP1A2 (e.g., cimetidine, fluvoxamine) or induce CYP1A2 (e.g., omeprazole) (Note: Subjects already on these agents may be enrolled, but must remain on stable doses of the agents from (Visit 1) 14 days prior to Baseline to the end of the study.
* Current hallucinations
* History of disabling hallucinations or hallucinations in past requiring treatment
* Mini-Mental status examination score < 25 on a scale of 30
* Orthostatic hypotension >30 systolic drop and >20 diastolic drop
* On cholinesterase inhibitors or memantine
* Troublesome edema due to any reason
* Epworth sleepiness scale >8
* Another primary sleep disorder (e.g. obstructive sleep apnea, narcolepsy)
* Secondary causes of RLS (iron deficiency, renal failure)
* Unstable medical conditions as determined by the investigator
* Inadequately managed depression (patient on antidepressants must be on stable dose for 4 weeks prior to enrollment)
* Other stable medical conditions which may interfere with patient evaluation
* Female who is pregnant or lactating
* Use of an investigational drug within the last 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-05; Primary Completion 2007-09 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
CGI-S/CGI-I: (Visits 1, 2, and 4) | 5 min
IRLS: (Visits 1, 2, and 4) | 5 min
Epworth Sleepiness Scale: (Visits 1, 2, and 4) | 5 min
ECG: An "ECG" or "electrocardiogram" is a test that measures the electrical activity of the heart. (Visits 1, 2, and 4) | 5 min

CONTACTS AND LOCATIONS:
Overall Officials: Kapil D Sethi, MD, Principal Investigator — Augusta University
Locations (1):
- Medical College of Georgia, Augusta, Georgia, United States